CLINICAL TRIAL: NCT05545072
Title: A Randomized, 52-week Treatment Double-blind, Placebo-controlled Efficacy and Safety Study of Dupilumab 300 mg Every Other Week After Endoscopic Sinus Surgery in Patients With Allergic Fungal Rhinosinusitis (AFRS) on a Background Therapy With Intranasal Corticosteroid Spray
Brief Title: Add-on Dupilumab for AFRS as Postoperative Therapy (ADAPT)
Acronym: ADAPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to funding ending.
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Joshua M. Levy, Adjunct Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000090
Record Dates: First submitted 2022-08-31; First posted 2022-09-19 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Allergic Fungal Rhinosinusitis
MeSH Terms: conditions — Allergic Fungal Sinusitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded, placebo-controlled, parallel-group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): Participants receiving dupilumab for 52 weeks following surgery for allergic fungal rhinosinusitis (AFRS).
  Interventions: Drug: Dupilumab; Drug: Intranasal Corticosteroid Sprays (INCS)
- Placebo (Placebo Comparator): Participants receiving a placebo to match dupilumab for 52 weeks following surgery for allergic fungal rhinosinusitis (AFRS).
  Interventions: Drug: Placebo; Drug: Intranasal Corticosteroid Sprays (INCS)

INTERVENTIONS:
Drug: Dupilumab — Dupilumab will be administered subcutaneously at a dose of 300 milligrams (mg) in a 2 milliliter (mL) solution every 2 weeks until the end of treatment (EOT) at Week 52. Participants will receive a total of 26 doses.
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Placebo — A placebo to match dupilumab will be administered subcutaneously every 2 weeks until the end of treatment (EOT) at Week 52. Participants will receive a total of 26 doses.
  Arms: Placebo
Drug: Intranasal Corticosteroid Sprays (INCS) — All participants will undergo standardized background therapy with intranasal corticosteroid sprays (INCS) per standard of care (SoC). This will continue throughout the entire study. Participants either receive fluticasone propionate or mometasone furoate.

SUMMARY:
The purpose of this study is to find a more effective treatment for allergic fungal rhinosinusitis (AFRS). Most people suffering from nasal polyps have elevated levels of white blood cells called eosinophils that are involved in inflammation of the air passages. Despite appropriate treatment with oral/topical corticosteroids, saline irrigations, and surgery, nasal polyps return frequently within months of surgery. Participants will be administered a placebo or dupilumab every two weeks for 52 weeks.

DETAILED DESCRIPTION:
Allergic fungal rhinosinusitis (AFRS) is a severe form of eosinophilic nasal polyposis with critically inadequate treatment options for the 10% of chronic rhinosinusitis subjects affected by the disease. Occlusive eosinophilic mucus and severe nasal polyposis present in early adulthood, with an unrelenting course marked by sinus expansion and pressure-induced dehiscence of the surrounding orbit and skull base. Despite appropriate therapies with oral/topical corticosteroids, saline irrigations, and comprehensive sinus surgery, nasal polyps aggressively recur, frequently within months of surgery. Medical options beyond topical and systemic steroids are limited. Neither antifungal nor allergen immunotherapy is beneficial. Due to persistent sinonasal inflammation, patients with AFRS receive an average of three corticosteroid bursts per year and revision sinus surgery every 42 months.

Certain proteins made by the body, called interleukins, appear to play a major role in the survival and activation of eosinophils. Antibodies are proteins naturally produced by your body that find foreign substances, such as bacteria, fungi, viruses, and other substances that enter your body and make them inactive. Dupilumab is an antibody made in the laboratory that has been made to block specific interleukins from activating the eosinophils. This research is being done to find out if the medication dupilumab is effective and safe when used to treat patients with AFRS following recommended sinus surgery. Dupilumab is already approved for the treatment of atopic dermatitis, asthma, and chronic rhinosinusitis with nasal polyposis (CRSwNP); however, it is not approved to treat AFRS.

Patients who meet the eligibility criteria will be enrolled in this randomized, double-blind study and will go through four periods: a run-in period, surgery period, randomized treatment period, and post-treatment period. During the run-in period, patients will perform twice daily saline irrigations followed by intranasal corticosteroid spray (INCS) for 2 to 6 weeks before planned sinus surgery. Saline irrigations/INCS and sinus surgery will be completed by the standard of care (SoC). Patients who continue to meet eligibility criteria following surgery will be randomized to receive a placebo or dupilumab subcutaneously every 2 weeks. Participants will receive 26 doses of the investigational medical product (IMP), via either study personnel or home administration, to maintain a 2-week treatment schedule. Participants will receive IMP directly from the central pharmacy, with compliance assessments via reminder text messages on the day of each scheduled home administration, as well as monthly phone calls and injection device collection at recurring 3-month study visits. Participants will then be monitored on daily saline irrigation and INCS spray for 12 weeks to evaluate potential disease recurrence after discontinuation of IMP. An end-of-study visit will be conducted 12 weeks after the treatment period at Week 64.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Patients aged >18 years at the time of signing the informed consent form (ICF)
* Patients with nasal polyps in the setting of suspected AFRS and electing to undergo comprehensive sinus surgery per established criteria

  * Diagnosis of nasal polyps by consensus criteria
  * Failure of appropriate medical therapy, including topical intranasal corticosteroid (spray or irrigation) > 8 weeks duration, systemic corticosteroid trial of 1-3 weeks duration, and nasal saline irrigation of > 4 weeks duration
  * A minimum SNOT-22 score of 20 at the time of enrollment
  * A minimum CT Lund-MacKay score of > 1 at the time of enrollment
* Suspected AFRS based on Bent and Kuhn criteria

  * Patients meet 3/5 criteria at the time of enrollment and 5/5 criteria at time of randomization: environmental atopy by skin or serum testing, nasal polyposis, characteristic CT findings, eosinophilic mucous, fungal identification on histopathology

Exclusion Criteria:

* Patients who have undergone nasal or sinus surgery within 3 months prior to enrollment
* Patients with conditions or comorbid disease findings that exclude nasal endoscopy for evaluation of primary outcomes, such as current rhinitis medicamentosa, nasal cavity tumors, occlusive septal deviation following surgery
* Clinically important comorbidities that may confound the interpretation of clinical efficacy, including aspirin-exacerbated respiratory disease, cystic fibrosis, primary ciliary dyskinesia, Hereditary Hemorrhagic Telangiectasia, antrochoanal polyposis, non-asthma eosinophilic disease (such as bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome), granulomatosis with polyangiitis, any corticosteroid-dependent condition
* A comorbid health disorder that is not medically controlled in the opinion of the Investigator, and has the potential to: affect the safety of the subject throughout the study, impede the subject's ability to complete the duration of the study, influence the primary or secondary outcomes of the study
* Patient experiencing a symptomatic asthma exacerbation requiring systemic corticosteroids or hospitalization (>24 hours) within 4 weeks of randomization
* Infection requiring systemic antibiotics within 4 weeks of randomization (parenteral and/or oral antibiotics associated with surgery are allowed)
* Medical contraindication to receiving dupilumab: known hypersensitivity to dupilumab or any of its excipients, live vaccine administration within 30 days of randomization or during the study period, known helminth infection
* Unable to tolerate sinonasal irrigations
* Pregnancy, current lactation, or lack of effective contraception plan, as determined by the site investigator
* Initiation of allergen immunotherapy within 3 months prior to randomization or a plan to begin therapy or change its dose during the study period
* Immunosuppressive medication within 3 months prior to randomization and during the study period from randomization through the end of the study
* Receipt of any marketed or investigational biologic products (monoclonal or polyclonal antibody) within 6 months or 5 half-lives, whichever is longer, prior to randomization during the study period
* Previous use of dupilumab
* Receipt of immunoglobulin or blood products within 30 days prior to randomization
* Receipt of any investigational drug within 30 days or 5 half-lives, whichever is longer prior to randomization
* Scheduled systemic corticosteroid treatment during the study period (standardized corticosteroid taper associated with planned surgery is allowed)
* Receipt of leukotriene antagonists or modifiers for subjects who were not on a stable dose for > 30 days prior to randomization
* Concurrent enrollment in another investigational drug trial during the study period
* Patient involvement in the planning or conduct of the study
* Investigator assessment that the subject is unlikely to comply with study procedures
* Prior randomization in the present study
* Unable to undergo sinus surgery due to comorbid medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Levy, MD, MPH, MSc, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Hospital Midtown-Otolaryngology, Atlanta, Georgia
  - Ambulatory Surgery Center - Emory University Hospital, Atlanta, Georgia
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share individual participant data that underline the results reported in the article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The investigators will share de-identified data beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to joshua.levy2@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were planned for recruitment from three locations in the USA: the University of Texas Health Science Center at Houston, in Houston, Texas, and Emory University Hospital Midtown and Emory University Hospital in Atlanta, Georgia. Participant enrollment began October 26, 2023, and the final study visit occurred July 10, 2024. The University of Texas Health Science Center at Houston was not activated as a site, and all participants were recruited at the Emory site.
Groups:
- Dupilumab: Participants receiving dupilumab for 52 weeks following surgery for allergic fungal rhinosinusitis (AFRS).
  Dupilumab: Dupilumab will be administered subcutaneously at a dose of 300 milligrams (mg) in a 2 milliliter (mL) solution every 2 weeks until the end of treatment (EOT) at Week 52. Participants will receive a total of 26 doses.
  Intranasal Corticosteroid Sprays (INCS): All participants will undergo standardized background therapy with intranasal corticosteroid sprays (INCS) per standard of care (SoC). This will be continued throughout the entire study. Participants either receive fluticasone propionate or mometasone furoate.
- Placebo: Participants receiving a placebo to match dupilumab for 52 weeks following surgery for allergic fungal rhinosinusitis (AFRS).
  Placebo: A placebo to match dupilumab will be administered subcutaneously every 2 weeks until the end of treatment (EOT) at Week 52. Participants will receive a total of 26 doses.
  Intranasal Corticosteroid Sprays (INCS): All participants will undergo standardized background therapy with intranasal corticosteroid sprays (INCS) per standard of care (SoC). This will be continued throughout the entire study. Participants either receive fluticasone propionate or mometasone furoate.
Period: Overall Study
Arm/Group | Dupilumab | Placebo
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study ended prematurely due to funding | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dupilumab | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Modified Lund-Kennedy (mLK) Score
Description: The efficacy of dupilumab in controlling sinonasal inflammation and preventing nasal polyp recurrence after complete sinus surgery for allergic fungal rhinosinusitis (AFRS) is assessed by using the modified Lund-Kennedy score. The modified Lund-Kennedy score (mLK) is a validated measure of sinonasal inflammation, as evaluated by means of nasal endoscopy. The composite score ranges from 0 to 12, with an increasing score representing worsening inflammation among three separate findings (Nasal polyps, Discharge, Edema). Each finding is rated from 0 (absent) to 2 (severe). A ≥ 2-point increase from baseline total postoperative score represents a clinically significant worsening of sinonasal inflammation.
Time Frame: Baseline and End of Treatment at Week 52
Population: Data are not available for the calculation of the mLK score as the study was terminated before central reader scoring of the nasal endoscopy.
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of Oral/Topical Corticosteroid Utilization Per Participant
Description: The number of participants who, during study treatment and off-treatment follow-up, based on clinical evaluation, present worsening signs and/or symptoms and are started on oral corticosteroids rescue treatment.
Time Frame: Baseline and End of Treatment at Week 52
Population: Participants were unable to complete the study visits as scheduled at 52 weeks due to the premature termination of the study. Data is reported up to the time point completed by all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Baseline | 3 | 2
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 0 | 0
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Prevalence of Revision Sinus Surgery for Recurrent Nasal Polyps, and Comparison of Survival Curves
Description: Documentation of the number of revision sinus surgery per participant, that are deemed clinically necessary for the treatment of an acute exacerbation of chronic rhinosinusitis (AECRS)
Time Frame: Up to End of Treatment at Week 52
Measure: Mean (Standard Deviation); unit: Revision Surgeries per participant
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Revision Surgeries per participant | 0 (0) | 0 (0)

4. Secondary Outcome: Endoscopic Nasal Polyp Score (NPS)
Description: NPS is a physician-reported tool to grade the extent/severity of nasal polyps based on evaluation by nasal endoscopy. Each nostril is scored on a scale of 0 (no polyps visible) to 4 (massive polyposis completely obstructing the nasal cavity), with the total score being the sum of left and right nostril scores (range: 0-8). The total NPS is the sum of scores from the right and left nostrils.
Time Frame: Baseline and End of Treatment at Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline | 4.33 (0.47) | 5 (1)
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 1 (0) | 0 (0)
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 2 (0) |
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Predicted Forced Vital Capacity (%FVC) Following Sinus Surgery in the Subgroup of Participants With Asthma (~25%)
Description: Spirometry is a common office test used to assess how well the participant's lungs work by measuring how much air the participant inhales, how much the participant exhales, and how quickly the participant exhales. Forced vital capacity (FVC) refers to the maximal volume of air that can be expired following maximum inspiration. It is the total of tidal volume, inspiratory reserve volume, and expiratory reserve volume. The percent FVC is the FVC compared to a predicted FVC based on age, sex, and height.
Time Frame: Baseline and End of Treatment at Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: %FVC
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 2 | 1
%FVC
  Baseline | 107 (3) | 104 (0)
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Following Sinus Surgery in the Subgroup of Participants With Asthma (~25%)
Description: Forced expiratory volume in one second (FEV1) is measured during a spirometry test, also known as a pulmonary function test, which involves forcefully breathing out into a mouthpiece connected to a spirometer machine. FEV1 is the amount of air forced from the lungs in one second.
Time Frame: Baseline and End of Treatment at Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 2 | 1
Liter
  Baseline | 3.55 (0.76) | 2.80 (0)
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Forced Vital Capacity (FVC) Following Sinus Surgery in the Subgroup of Participants With Asthma (~25%)
Description: Forced vital capacity (FVC) is measured during a spirometry test, also known as a pulmonary function test, which involves forcefully breathing out into a mouthpiece connected to a spirometer machine. FVC is the total amount of air exhaled during the FEV test.
Time Frame: Baseline and End of Treatment at Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
liter
  Baseline: number analyzed (Participants) | 2 | 1
  Baseline | 4.67 (1.07) | 3.53 (0)
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: FEV1/FVC Ratio Following Sinus Surgery in the Subgroup of Participants With Asthma (~25%)
Description: The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. The normal value for this ratio is above 0.75-85, though this is age-dependent, values less than 0.70 are suggestive of airflow limitation with an obstructive pattern.
Time Frame: Baseline and End of Treatment at Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: FEV1/FVC
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
FEV1/FVC
  Baseline: number analyzed (Participants) | 2 | 1
  Baseline | 0.76 (0.01) | 0.79 (0)
  End of Treatment at Week 52: number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in the Modified Lund-Kennedy (mLK) Radiologic Score
Description: The mLK Radiologic scoring system assigns a value of 0, 1, or 2 to each of the following sinuses: maxillary, anterior ethmoid, posterior ethmoid, frontal, and sphenoid. Score assignments are 0 if the sinus is totally patent, 1 if the sinus is partially opacified, and 2 if the sinus is completely opacified. The osteomeatal complex is scored either 0 if not occluded or 2 if occluded. The maximum score for each side is thus 12, with a total score determined out of 24. Baseline Lund- MacKay (LM) scores will be counted as zero in accordance with recent sinus surgery.
Time Frame: 52 weeks and 64 weeks
Population: Data for the calculation of the mLK score are not available, as the study was terminated prematurely before participants were able to complete the scheduled study visits at weeks 52 and 64.
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Endoscopic Nasal Polyp Score (NPS)
Description: Endoscopic nasal polyp score is determined by the treating Investigator. Unlike prior studies of dupilumab in nasal polyps, researchers will separately record the Nasal Polyp Score for each side, with a maximum unilateral score of 4 (massive polyposis completely obstructing the nasal cavity). This is appropriate for monitoring efficacy in AFRS, as a subgroup of participants may present with unilateral disease.
Time Frame: 52 weeks and 64 weeks
Population: Participants were unable to complete the study visits as scheduled at 52 and 64 weeks due to the premature termination of the study.
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: The 22-item Sinonasal Outcomes Test (SNOT-22) Score
Description: The SNOT-22 score is a validated disease-specific questionnaire quantifying the quality of life among participants with chronic rhinosinusitis. The individual question scores range from 0 (no problem) to 4 (as bad as it can be) among 22 separate questions. Scoring 0 to 110. Higher scores = more severe symptoms and poorer quality of life.
Time Frame: 52 weeks and 64 weeks
Population: Participants were unable to complete the study visits as scheduled at 52 and 64 weeks due to the premature termination of the study. Data is reported up to the time point completed by all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale
  Baseline | 37 (14.73) | 17 (5.66)
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 13 (0) | 2 (0)
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 12 (0) |
  52 Weeks: number analyzed (Participants) | 0 | 0
  64 weeks: number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Asthma Control Questionnaire (ACQ) Score Among Participants With Asthma
Description: The Asthma Control Questionnaire (ACQ) is a validated, self-administered survey used to assess a participants' perception of disease control over the preceding week using Likert scale responses with a range of 0 (well controlled) to 6 (extremely poorly controlled). The ACQ consists of 7 items surveying the frequency of asthma related symptoms, the need for rescue medications, and perceived control of disease. The items are equally weighted and the ACQ score is the mean of the 7 items. Total scores range from 0 to 6 with lower scores indicating better control of asthma symptoms. A score change of 0.5 on the 7-point scale has previously been defined as the Minimal Important Difference (MID).
Time Frame: 52 weeks and 64 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Score on a scale
  Baseline: number analyzed (Participants) | 2 | 1
  Baseline | 5.5 (0.5) | 6 (0)
  52 weeks: number analyzed (Participants) | 0 | 0
  64 weeks: number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Prevalence of Oral/Topical Corticosteroid Utilization Per Treatment Cohort
Description: The number of participants who, during study treatment and off-treatment follow-up, based on clinical evaluation, have to continue on oral corticosteroid rescue treatment due to worsening signs and/or symptoms.
Time Frame: 52 weeks and 64 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Baseline | 0 | 0
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 0 | 0
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |
  Week 54: number analyzed (Participants) | 0 | 0
  Week 64: number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Incidence of Oral/Topical Antibiotic Utilization Per Participant
Description: The number of participants who, during study treatment and off-treatment follow-up, based on clinical evaluation, present worsening signs and/or symptoms and are started on oral/topical antibiotic rescue treatment.
Time Frame: 52 weeks and 64 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Baseline | 0 | 0
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 0 | 0
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |
  Weeks 54: number analyzed (Participants) | 0 | 0
  Week 64: number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Prevalence of Oral/Topical Antibiotic Utilization Per Treatment Cohort
Description: The number of participants who, during study treatment and off-treatment follow-up, based on clinical evaluation, have to continue on oral/topical antibiotic rescue treatment due to worsening signs and/or symptoms.
Time Frame: 52 weeks and 64 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Baseline | 0 | 0
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12 | 0 | 0
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |
  Week 54: number analyzed (Participants) | 0 | 0
  Week 64: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at run-in (Week -6) and continued through the final assessment at Week 24 until the study premature termination.
Arm/Group | Dupilumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dupilumab (N=3) | Placebo (N=2)
Headache (Nervous system disorders) | 1 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2 | 2
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Other (General disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT05545072/Prot_SAP_000.pdf